CLINICAL TRIAL: NCT03976908
Title: Deep Brain Stimulation for Refractory Tinnitus
Brief Title: Deep Brain Stimulation for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL67027.068.18
Record Dates: First submitted 2019-03-07; First posted 2019-06-06 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Tinnitus
Keywords: Tinnitus; Deep Brain Stimulation
MeSH Terms: conditions — Tinnitus | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Clinical intervention study (double blind, randomized cross-over design). Two different stimulation paradigms will be investigated: ON and OFF stimulation.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ON-OFF (Experimental): Patients receive the same baseline, a 6 week period of stimulation ON (masked for both patient and investigator), one week of washout, a 6 week period of stimulation OFF (masked for both patient and investigator), one week of washout, a 6 month follow-up period of open-label stimulation ON.
  Interventions: Device: Deep Brain Stimulation
- OFF-ON (Experimental): Patients receive the same baseline, a 6 week period of stimulation OFF (masked for both patient and investigator), one week of washout, a 6 week period of stimulation ON (masked for both patient and investigator), one week of washout, a 6 month follow-up period of open-label stimulation ON.
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — High frequency deep brain stimulation in the medial geniculate body of the thalamus.

SUMMARY:
Tinnitus is the perception of a sound in the absence of an audible source. Currently up to 15% of the general population suffers chronically from tinnitus. The most severe degree of tinnitus ís experienced by 2.4% of the population and is associated with insomnia, depression; anxiety and even suicide. Up to date there is no effective standard therapy. Current therapies mostly focus on treating the distress caused by tinnitus instead of reducing the actual phantom sound. Nevertheless, many patients do not benefit from the current approaches and become severe and chronic tinnitus sufferers. In these patients neuromodulation-based treatments can be a promising option. Tinnitus perception is associated with many complex changes in several different brain structures. The general accepted hypothesis is that neuronal changes occur in both auditory and non-auditory brain structures, most often as a compensating mechanism on reduced input from the auditory nerve caused by cochlear hair cell damage. These central neuronal changes include an increase in spontaneous firing rate, synchronized activity, bursting activity and tonotopic reorganization. In high-frequency deep brain stimulation (DBS) a reversible lesion-like effect is mimicked. From findings in Parkinson's disease patients who also had tinnitus and were treated with DBS, it is known that stimulation can alter or even completely diminish perception of tinnitus. It can be expected that modulation of specific structures within the complex tinnitus pathways can disrupt pathological neuronal activity and thereby alter tinnitus perception or distress caused by this phantom sensation. The investigators found in animal studies that DBS in the central auditory pathway can indeed significantly decrease tinnitus-like behavior. In a questionnaire study the investigators found that around one-fifth of the patients would be reasonably willing to accept invasive treatments and one-fifth would be fully willing to undergo invasive treatment like DBS. Based on preclinical studies and human case studies, the investigators expect that DBS of the central auditory pathway will inhibit tinnitus perception and distress caused by this phantom sensation. Based on studies performed within Maastricht University Medical Center (MUMC), the investigators selected the medial geniculate body of the thalamus (MGB) as the most potential target to treat tinnitus with DBS.

ELIGIBILITY:
Inclusion Criteria:

* Medically refractory tinnitus. Patient does not respond to available tinnitus treatments (hearing aids, cognitive treatments) and is thoroughly evaluated by the multidisciplinary tinnitus team in MUMC. Thus patients do not respond to both of the following treatments (i.e. TQ is still ≥ 47):
* Hearing aids (except if hearing is normal)
* Evidence-based cognitive treatment in Hoensbroek (Cima et al., 2012) or a similar version of this treatment in the MUMC
* Minimum age 18 years, maximum age 69 years.
* Experiencing tinnitus which is:
* Not pulsatile
* Unilateral or bilateral
* Severe tinnitus (based on the TQ score ≥ 47)
* Chronic and stable (present > 2 years and stable > 1 year).
* Bilateral hearing of high tone Fletcher Index < 60 dB
* Willingness to participate in this study (informed consent)

Exclusion Criteria:

* Anatomic cause of tinnitus (e.g. vestibular schwannoma, tumour, middle-ear pathology)
* DSM-V psychiatric disorders, other than depression or anxiety disorder (such as bipolar disorder, dementia, addiction, personality disorders); diagnosed by a psychiatrist. A psychiatrist will screen the patients for this matter.
* Depression or anxiety disorder which was already present before tinnitus. A psychiatrist will screen the patients for this matter.
* Cognitive impairment (assessed with standard 'cognitive functioning battery test' questionnaires) or coping problems (CISS-21)
* Active ear diseases that needs further attention according to research team
* Pregnancy or breast-feeding
* Active suicide thoughts or attempts
* Underlying malignancies, whenever life expectancy is lower than 2 years
* Other implantable electronic devices that potentially could interfere with DBS, e.g. cochlear implants, auditory brainstem implants or cortical implants

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change over time of the score on the Tinnitus Functional Index | Week 1, week 20, week 26, week 33, week 60
  A validated questionnaire which assesses the impact of tinnitus on a patient measured on multiple time points to measure a change over time. The TFI score can range from 0-100, higher values indicate more tinnitus burden. When a patient scores 54 or higher the tinnitus is considered to be a major problem.

SECONDARY OUTCOMES:
VAS Loudness | Week 1, week 12, week 20, week 26, week 33, week 60
  on a scale from 0 (no tinnitus) to 10 (most severe tinnitus imaginable), subjects rate their tinnitus perception on loudness.
VAS Burden | Week 1, week 12, week 20, week 26, week 33, week 60
  on a scale from 0 (no tinnitus) to 10 (most severe tinnitus imaginable), subjects rate their tinnitus perception amount of discomfort.
15 word memory test | Week 1, week 27, week 34, week 60
  Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat. Another list of 15 unrelated words are given and the client must again repeat the original list of 15 words and then again after 30 minutes.
Boston naming test | Week 1, week 27, week 34, week 60
  The neurpsychologist shows the person each of the pictures, one at a time in the given order. The person is given 20 seconds to say what the drawing depicts.
Stroop Color and Word Test | Week 1, week 27, week 34, week 60
  This is a neuropsychological test used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect.
Trail Making Test | Week 1, week 27, week 34, week 60
  This is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy.
Semantic Verbal Fluency Test (Animals) | Week 1, week 27, week 34, week 60
  This is a test in which participants have to produce as many words as possible from a category, here animals.
Semantic Verbal Fluency Test (Jobs) | Week 1, week 27, week 34, week 60
  This is a test in which participants have to produce as many words as possible from a category, here jobs.
Phonemic Verbal Fluency Test (D) | Week 1, week 27, week 34, week 60
  This is a test in which participants have to produce as many words as possible from a category, here words starting with the letter D.
Phonemic Verbal Fluency Test (A) | Week 1, week 27, week 34, week 60
  This is a test in which participants have to produce as many words as possible from a category, here words starting with the letter A.
Phonemic Verbal Fluency Test (T) | Week 1, week 27, week 34, week 60
  This is a test in which participants have to produce as many words as possible from a category, here words starting with the letter T.
Quality of life Questionnaire | Week 1, week 27, week 34, week 60
  The Short Form (36) Health Survey (standard validated questionnaire)
Beck Depression Inventory II (BDI-II) | Week 1, week 60
  Validated questionnaire for depression.
Beck Anxiety Inventory (BAI) | Week 1, week 60
  Validated questionnaire for anxiety.
Hospital Anxiety and Depression Scale (HADS) | Week 1, week 60
  Validated questionnaire for anxiety and depression.
Audiometry | Week 1, week 14, week 27, week 34, week 60
  pure-tone and speech audiometry. These are the clinical standard audiometric tests.
Auditory Brainstem Response | Week 1, week 14, week 27, week 34, week 60
  Neurophysiological measure following standard protocols.
Electroencephalography (EEG) | Week 1, week 14, week 27, week 34, week 60
  Neurophysiological measure following standard protocols.
Local Field Potentials (LFP) | Week 12
  Neurophysiological measure following standard protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Janssen, Dr., Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] van Zwieten G, Devos JVP, Kotz SA, Ackermans L, Brinkmann P, Dauven L, George ELJ, Janssen AML, Kremer B, Leue C, Schwartze M, Temel Y, Smit JV, Janssen MLF. A Protocol to Investigate Deep Brain Stimulation for Refractory Tinnitus: From Rat Model to the Set-Up of a Human Pilot Study. Audiol Res. 2022 Dec 31;13(1):49-63. doi: 10.3390/audiolres13010005. PMID 36648926